CLINICAL TRIAL: NCT01970501
Title: GENETIC-AF - A Genotype-Directed Comparative Effectiveness Trial of Bucindolol and Toprol-XL for Prevention of Symptomatic Atrial Fibrillation/Atrial Flutter in Patients With Heart Failure
Brief Title: Genetically Targeted Therapy for the Prevention of Symptomatic Atrial Fibrillation in Patients With Heart Failure
Acronym: GENETIC-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-CLIN-303
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Current or Recent History of Atrial Fibrillation
Keywords: atrial fibrillation; atrial flutter; heart failure; reduced left ventricle ejection fraction; electrical cardioversion; GENETIC-AF; Medtronic; bucindolol; pharmacogenetic; ARCA; Toprol; Toprol-XL; Metoprolol; Metoprolol succinate
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Heart Failure | interventions — bucindolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bucindolol hydrochloride (Experimental): bucindolol hydrochloride (bucindolol)
  Participants were randomized (1:1) to blinded treatment with bucindolol or metoprolol and titrated weekly to target doses of 50 mg twice daily (BID; < 75 kg) or 100 mg BID (≥ 75 kg) for bucindolol or 200 mg once daily (QD) for metoprolol. 84% of bucindolol participants attained target dose and 72% of metoprolol participants attained target dose.
  The lowest starting dose of bucindolol was 6.25 mg BID with weekly dose titrations to the weight-based target dose or to the maximum tolerated dose. The starting dose assigned was based on the patient's beta-blocker treatment prior to randomization. Capsules for titration were available in the following dosage strengths to be taken twice daily (with or without food): 6.25mg, 12.5mg, 25mg, 50mg, and 100mg.
  Interventions: Drug: bucindolol hydrochloride
- metoprolol succinate (Active Comparator): metoprolol succinate (Toprol-XL)
  Participants were randomized (1:1) to blinded treatment with bucindolol or metoprolol and titrated weekly to target doses of 50 mg twice daily (BID; < 75 kg) or 100 mg BID (≥ 75 kg) for bucindolol or 200 mg once daily (QD) for metoprolol. 84% of bucindolol participants attained target dose and 72% of metoprolol participants attained target dose.
  The lowest starting dose of metoprolol was 25 mg QD with weekly dose titrations to the target dose or to the maximum tolerated dose. The starting dose assigned was based upon the patient's beta-blocker treatment prior to randomization. Capsules for titration were available in the following dosage strengths to be taken twice daily (with or without food): 25mg, 50mg, 100mg, 200mg and/or matching placebo oral capsule to maintain blinded dosing.
  Interventions: Drug: metoprolol succinate; Other: Placebo oral capsule

INTERVENTIONS:
Drug: bucindolol hydrochloride
  Other Names: bucindolol
  Arms: bucindolol hydrochloride
Drug: metoprolol succinate
  Other Names: Toprol-XL; metoprolol
  Arms: metoprolol succinate
Other: Placebo oral capsule
  Other Names: placebo
  Arms: metoprolol succinate

SUMMARY:
This study is being done to compare the effects of bucindolol hydrochloride (bucindolol) to metoprolol succinate (Toprol-XL) on the recurrence of symptomatic atrial fibrillation/atrial flutter in patients with heart failure who have a specific genotype for the beta-1 adrenergic receptor.

DETAILED DESCRIPTION:
The goal of the GENETIC-AF trial is to demonstrate the superiority of pharmacogenetically targeted bucindolol compared to metoprolol for the prevention of symptomatic atrial fibrillation or atrial flutter in a genotype-defined population with heart failure and/or reduced left ventricular ejection fraction at high risk of atrial fibrillation/atrial flutter recurrence.

ELIGIBILITY:
Key Inclusion Criteria:

* Must weigh at least 40 kg
* Possess the β1389 Arg/Arg genotype
* Left Ventricular Ejection Fraction (LVEF) < 0.50 assessed within 12 months prior to Screening
* At least one episode of symptomatic paroxysmal or persistent AF within 180 days of Screening
* Clinically appropriate for electrical cardioversion (ECV) if AF/AFL is present after study drug initiation
* Receiving appropriate anticoagulation therapy prior to Randomization

Key Exclusion Criteria:

* NYHA Class IV symptoms at the time of Randomization
* Significant fluid overload at Randomization
* Permanent AF at Screening
* More than two previous ECV within 6 months of Randomization or if the most recent ECV failed to produce SR
* Presence of an LVAD, or likely to requirement LVAD placement within 6 months of Randomization
* History of a successful atrioventricular (AV) node ablation
* History of an AF/AFL ablation within 30 days of Randomization
* Evidence of an appropriate firing of an implanted cardioverter-defibrillator (ICD) device for ventricular tachycardia (VT) or ventricular fibrillation (VF) within 90 days of Randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Piccini, MD, Principal Investigator — Duke University; Michael Bristow, MD,PhD, Study Director — ARCA Biopharma, Inc.
Locations (97):
- United States (48):
  - ARCA Clinical Research Site #157, Anchorage, Alaska
  - ARCA Clinical Research Site #383, Phoenix, Arizona
  - ARCA Clinical Research Site #385, Phoenix, Arizona
  - ARCA Clinical Research Site #381, East Palo Alto, California
  - ARCA Clinical Research Site #186, Loma Linda, California
  - ARCA Clinical Research Site #320, Pasadena, California
  - ARCA Clinical Research Site #390, Stanford, California
  - ARCA Clinical Research Site #153, Aurora, Colorado
  - ARCA Clinical Research Site #380, Denver, Colorado
  - ARCA Clinical Research Site #195, Miami, Florida
  - ARCA Clinical Research Site #184, Tampa, Florida
  - ARCA Clinical Research Site #351, Athens, Georgia
  - ARCA Clinical Research Site #389, Atlanta, Georgia
  - ARCA Clinical Research Site #342, Oakbrook Terrace, Illinois
  - ARCA Clinical Research Site #303, Hammond, Indiana
  - ARCA Clinical Research Site #388, Iowa City, Iowa
  - ARCA Clinical Site #396, New Orleans, Louisiana
  - ARCA Clinical Research Site #398, Baltimore, Maryland
  - ARCA Clinical Research Site #127, Ypsilanti, Michigan
  - ARCA Clinical Research Site #156, Minneapolis, Minnesota
  - ARCA Clinical Research Site #174, Saint Paul, Minnesota
  - ARCA Clinical Research Site #108, St Louis, Missouri
  - ARCA Clinical Research Site #201, St Louis, Missouri
  - ARCA Clinical Research Site #152, Lincoln, Nebraska
  - ARCA Clinical Research Site #161, Elmer, New Jersey
  - ARCA Clinical Research Site #202, Hillsborough, New Jersey
  - ARCA Clinical Research Site # 179, Albany, New York
  - ARCA Clinical Research Site #397, New York, New York
  - ARCA Clinical Research Site #181, Durham, North Carolina
  - ARCA Clinical Research Site #349, Greensboro, North Carolina
  - ARCA Clinical Research Site #173, Akron, Ohio
  - ARCA Clinical Research Site #392, Cincinnati, Ohio
  - ARCA Clinical Research Site #322, Cleveland, Ohio
  - ARCA Clinical Research Site #151, Columbus, Ohio
  - ARCA Clinical Research Site #399, Oklahoma City, Oklahoma
  - ARCA Clinical Research Site #115, Portland, Oregon
  - ARCA Clinical Research Site # 189, Hershey, Pennsylvania
  - ARCA Clinical Research Site #109, Lancaster, Pennsylvania
  - ARCA Clinical Research Site #133, Philadelphia, Pennsylvania
  - ARCA Clinical Site #393, Germantown, Tennessee
  - ARCA Clinical Research Site #198, Jackson, Tennessee
  - ARCA Clinical Research Site #387, Dallas, Texas
  - ARCA Clinical Research Site #379, Salt Lake City, Utah
  - ARCA Clinical Site #391, Charlottesville, Virginia
  - ARCA Clinical Research Site #386, Falls Church, Virginia
  - ARCA Clinical Research Site #200, Manassas, Virginia
  - ARCA Research Site #131, Norfolk, Virginia
  - ARCA Clinical Research Site #196, Puyallup, Washington
- Canada (18):
  - ARCA Clinical Research Site #612, Calgary, Alberta
  - ARCA Clinical Research Site #624, Vancouver, British Columbia
  - ARCA Clinical Research Site #611, Cambridge, Ontario
  - ARCA Clinical Research Site #621, Cambridge, Ontario
  - ARCA Clinical Research Site #601, Hamilton, Ontario
  - ARCA Clinical Research Site #609, London, Ontario
  - ARCA Clinical Research Site #623, Newmarket, Ontario
  - ARCA Clinical Research Site #618, Oshawa, Ontario
  - ARCA Clinical Research Site #613, Ottawa, Ontario
  - ARCA Clinical Research Site #619, Toronto, Ontario
  - ARCA Clinical Research Site #616, Waterloo, Ontario
  - ARCA Clinical Research Site #614, Montreal, Quebec
  - ARCA Clinical Research Site #607, Montreal, Quebec
  - ARCA Clinical Research Site #603, Montreal, Quebec
  - ARCA Clinical Research Site #625, Saint-Jérôme, Quebec
  - ARCA Clinical Research Site #602, Sherbrooke, Quebec
  - ARCA Clinical Research Site #626, Trois-Rivières, Quebec
  - ARCA Clinical Research Site #615, Québec
- Hungary (9):
  - ARCA Clinical Research Site #726, Budapest
  - ARCA Clinical Research Site #727, Budapest
  - ARCA Clinical Research Site #728, Budapest
  - ARCA Clinical Research Site #729, Budapest
  - ARCA Clinical Research Site #733, Debrecen
  - ARCA Clinical Research Site #732, Kaposvár
  - ARCA Clinical Research Site #730, Pécs
  - ARCA Clinical Research Site #731, Szeged
  - ARCA Clinical Research Site #734, Szolnok
- Netherlands (9):
  - ARCA Clinical Research Site #781, Capelle aan den IJssel
  - ARCA Clinical Research Site #779, Gorinchem
  - ARCA Clinical Research Site #776, Groningen
  - ARCA Clinical Research Site #780, Helmond
  - ARCA Clinical Research Site #782, Leiderdorp
  - ARCA Clinical Research Site #786, Roosendaal
  - ARCA Clinical Research Site #777, Sneek
  - ARCA Clinical Research Site #783, Stadskanaal
  - ARCA Clinical Research Site #784, Tiel
- Poland (8):
  - ARCA Clinical Research Site #752, Bialystok
  - ARCA Clinical Research Site #757, Gdansk
  - ARCA Clinical Research Site #753, Krakow
  - ARCA Clinical Research Site #755, Lodz
  - ARCA Clinical Research Site #751, Lodz
  - ARCA Clinical Research Site #758, Lublin
  - ARCA Clinical Research Site #754, Warsaw
  - ARCA Clinical Research Site #756, Wroclaw
- Serbia (5):
  - ARCA Clinical Research Site #807, Belgrade
  - ARCA Clinical Research Site #806, Belgrade
  - ARCA Clinical Research Site #801, Kragujevac
  - ARCA Clinical Research Site #804, Niš
  - ARCA Clinical Research Site #805, Niš

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liggett SB, Mialet-Perez J, Thaneemit-Chen S, Weber SA, Greene SM, Hodne D, Nelson B, Morrison J, Domanski MJ, Wagoner LE, Abraham WT, Anderson JL, Carlquist JF, Krause-Steinrauf HJ, Lazzeroni LC, Port JD, Lavori PW, Bristow MR. A polymorphism within a conserved beta(1)-adrenergic receptor motif alters cardiac function and beta-blocker response in human heart failure. Proc Natl Acad Sci U S A. 2006 Jul 25;103(30):11288-93. doi: 10.1073/pnas.0509937103. Epub 2006 Jul 14. PMID 16844790
- [Background] O'Connor CM, Fiuzat M, Carson PE, Anand IS, Plehn JF, Gottlieb SS, Silver MA, Lindenfeld J, Miller AB, White M, Walsh R, Nelson P, Medway A, Davis G, Robertson AD, Port JD, Carr J, Murphy GA, Lazzeroni LC, Abraham WT, Liggett SB, Bristow MR. Combinatorial pharmacogenetic interactions of bucindolol and beta1, alpha2C adrenergic receptor polymorphisms. PLoS One. 2012;7(10):e44324. doi: 10.1371/journal.pone.0044324. Epub 2012 Oct 10. PMID 23071495
- [Background] Aleong RG, Sauer WH, Davis G, Murphy GA, Port JD, Anand IS, Fiuzat M, O'Connor CM, Abraham WT, Liggett SB, Bristow MR. Prevention of atrial fibrillation by bucindolol is dependent on the beta(1)389 Arg/Gly adrenergic receptor polymorphism. JACC Heart Fail. 2013 Aug;1(4):338-344. doi: 10.1016/j.jchf.2013.04.002. PMID 24159564
- [Background] Kao DP, Davis G, Aleong R, O'Connor CM, Fiuzat M, Carson PE, Anand IS, Plehn JF, Gottlieb SS, Silver MA, Lindenfeld J, Miller AB, White M, Murphy GA, Sauer W, Bristow MR. Effect of bucindolol on heart failure outcomes and heart rate response in patients with reduced ejection fraction heart failure and atrial fibrillation. Eur J Heart Fail. 2013 Mar;15(3):324-33. doi: 10.1093/eurjhf/hfs181. Epub 2012 Dec 7. PMID 23223178
- [Derived] Carroll IA, Piccini JP, Steinberg BA, Tzou WS, Richards JC, DeMets DL, Bristow MR. Symptoms Burden as a Clinical Outcomes Assessment in Heart Failure Patients With Atrial Fibrillation. JACC Heart Fail. 2025 Apr;13(4):573-585. doi: 10.1016/j.jchf.2024.08.023. Epub 2024 Nov 20. PMID 39570238
- [Derived] Piccini JP, Dufton C, Carroll IA, Healey JS, Abraham WT, Khaykin Y, Aleong R, Krueger SK, Sauer WH, Wilton SB, Rienstra M, van Veldhuisen DJ, Anand IS, White M, Camm AJ, Ziegler PD, Marshall D, Bristow MR, Connolly SJ; Genotype-Directed Comparative Effectiveness Trial of Bucindolol and Toprol-XL for Prevention of Atrial Fibrillation/Atrial Flutter in Patients with Heart Failure Trial Investigators*. Bucindolol Decreases Atrial Fibrillation Burden in Patients With Heart Failure and the ADRB1 Arg389Arg Genotype. Circ Arrhythm Electrophysiol. 2021 Aug;14(8):e009591. doi: 10.1161/CIRCEP.120.009591. Epub 2021 Jul 16. PMID 34270905
- [Derived] Piccini JP, Connolly SJ, Abraham WT, Healey JS, Steinberg BA, Al-Khalidi HR, Dignacco P, van Veldhuisen DJ, Sauer WH, White M, Wilton SB, Anand IS, Dufton C, Marshall DA, Aleong RG, Davis GW, Clark RL, Emery LL, Bristow MR. A genotype-directed comparative effectiveness trial of Bucindolol and metoprolol succinate for prevention of symptomatic atrial fibrillation/atrial flutter in patients with heart failure: Rationale and design of the GENETIC-AF trial. Am Heart J. 2018 May;199:51-58. doi: 10.1016/j.ahj.2017.12.001. Epub 2017 Dec 6. PMID 29754666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment period began in Feb 2014 and the first participant screen was Apr 2014 and first randomization was Jun 2014. Recruitment continued through Jul 2017. Recruitment periods by country as follows:
  Canada: Mar 15 - Jul 17 Hungary: Sep 16 - Jun 17 Netherlands: May 1 - Jul 17 Poland: Jan 17 - Jul 17 Serbia: May 17 - Jun 17 United States: Feb 14 - Jul 17
Pre-assignment Details: During the drug lead in period, participants were uptitrated to target doses of each drug. Bucindolol target dose was 50 mg bid (subjects < 75 kg) or 100 mg bid (subjects >= 75 kg) or maximum tolerated dose. Metoprolol succinate target dose was 200 mg once daily or the maximum tolerated dose. Within each treatment arm, participants were combined for analysis.
Groups:
- Bucindolol Hydrochloride: Participants were randomized (1:1) to blinded treatment with bucindolol or metoprolol and titrated weekly to target doses of 50 mg twice daily (BID; < 75 kg) or 100 mg BID (≥ 75 kg) for bucindolol or 200 mg once daily (QD) for metoprolol. The starting dose of bucindolol was 6.25 mg BID with weekly dose titrations to the target dose or to the maximum tolerated dose. The bucindolol target dose varied based on the patient's weight on the day of randomization: patients < 75 kg receiving a target dose of 50 mg BID (100 mg daily) and patients > 75 kg receiving a target dose of 100 mg BID (200 mg daily).
  Capsules were available for titration in the following dosage strengths to be taken twice daily (with or without food): 6.25mg, 12.5mg, 25mg, 50mg, and 100mg.
- Metoprolol Succinate: metoprolol succinate (Toprol-XL)
  Participants were randomized (1:1) to blinded treatment with bucindolol or metoprolol and titrated weekly to target doses of 50 mg twice daily (BID; < 75 kg) or 100 mg BID (≥ 75 kg) for bucindolol or 200 mg once daily (QD) for metoprolol. The starting dose of bucindolol was 6.25 mg BID with weekly dose titrations to the target dose or to the maximum tolerated dose. The bucindolol target dose varied based on the patient's weight on the day of randomization: patients < 75 kg receiving a target dose of 50 mg BID (100 mg daily) and patients > 75 kg receiving a target dose of 100 mg BID (200 mg daily).
  Capsules were available for titration in the following dosage strengths to be taken twice daily (with or without food): 25mg, 50mg, 100mg, 200mg and/or matching placebo oral capsule to maintain blinded dosing.
Period: Overall Study
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
Started | 134 | 133
Randomization (Visit 2) (Blinding will be accomplished by providing study drug (i.e., bucindolol or metoprolol tablets) in capsules that are visually indistinguishable and provided in numbered kits. Only the numbers of the kits to be administered to a given patient, and not the identity of the study drug, will be provided to sites. Investigators, site personnel, and patients will not be informed of the blinded study drug assignment at the time of study completion.) | 134 | 133
Initial Dose Level 1 (Either Bucindolol 6.25mg BID or Metoprolol XL 25mg QD) | 35 | 45
Initial Dose Level 2 (Either Bucindolol 12.5 mg BID or Metoprolol XL 50 mg QD) | 45 | 38
Initial Dose Level 3 (Either Bucindolol 25 mg BID or Metoprolol XL 100 mg QD) | 51 | 45
Initial Dose Level 4 (Either Bucindolol 50 mg BID or Metoprolol XL 200 mg QD) | 3 | 5
Drug Lead-in Period (Bucindolol taken twice daily. Starting dose of 6.25 mg, 12.5 mg, 25 mg, or 50 mg bid depending upon pre-study beta-blocker dose. Sites instructed to uptitrate to target dose of 50 mg bid (subjects < 75 kg) or 100 mg bid (subjects >= 75 kg). Metoprolol succinate taken once per day and a placebo capsule taken once per day. Metoprolol succinate starting dose is 25 mg daily with dose titrations until 200 mg once daily or the maximum tolerated dose is achieved.) | 134 | 133
Attained Target Dose | 112 | 96
24-Week Follow Up Period (Sponsor requested that the last visit be between Aug-Dec 2017 and therefore a number of participants completed this arm prior to 24 week and are noted as sponsor or investigator initiated.) | 132 | 126
Treatment Extension Period (Sponsor requested that the last visit be between Aug-Dec 2017 and therefore a majority of participants were not enrolled in this treatment extension period.) | 77 | 64
Completed | 107 | 105
Not Completed | 27 | 28
Not completed — Discontinuation of study by sponsor | 16 | 14
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Adverse Event | 2 | 4
Not completed — Death | 1 | 3
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bucindolol Hydrochloride: bucindolol hydrochloride (bucindolol)
  Capsules are available in the following dosage strengths to be taken twice daily (with or without food): 6.25mg, 12.5mg, 25mg, 50mg, and 100mg.
  bucindolol hydrochloride
- Metoprolol Succinate: metoprolol succinate (Toprol-XL)
  Capsules are available in the following dosage strengths to be taken twice daily (with or without food): 25mg, 50mg, 100mg, 200mg and/or matching placebo oral capsule to maintain blinded dosing.
  metoprolol succinate
  Placebo oral capsule
- Total: Total of all reporting groups
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate | Total
Number analyzed (Participants) | 134 | 133 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 53 | 109
  >=65 years | 78 | 80 | 158
Age, Continuous [Mean (Full Range); unit: years] | 65 [40 to 86] | 65 [35 to 89] | 65 [35 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 111 | 108 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 129 | 128 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 27 | 59
  Netherlands | 2 | 2 | 4
  Hungary | 18 | 15 | 33
  United States | 60 | 67 | 127
  Poland | 13 | 10 | 23
  Serbia | 9 | 12 | 21
New York Heart Association (NYHA) Functional Class at screen [Count of Participants; unit: Participants] — Class I: No limitation of physical activity. Class II(Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea. Class III(Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV(Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
  Participants
    NYHA I | 40 | 35 | 75
    NYHA II | 80 | 72 | 152
    NYHA III | 14 | 26 | 40
    NYHA IV | 0 | 0 | 0
Ischemic Heart Failure [Count of Participants; unit: Participants] | 42 | 44 | 86
Non-Ischemic Heart Failure [Count of Participants; unit: Participants] | 92 | 89 | 181
Average Left Ventricular Ejection Fraction (LVEF) (%) [Mean (Full Range); unit: %] — A healthy (normal) ejection fraction is between 50-70%. Borderline ejection fraction is between 41-49% and reduced ejection fraction is <40%, indicating the heart is not adequately pumping blood to the body.
  % | 36 [10 to 49] | 36 [10 to 49] | 36 [10 to 49]
Rhythm at randomization [Count of Participants; unit: Participants]
  Atrial Fibrillation | 66 | 69 | 135
  Sinus Rhythm | 68 | 64 | 132
Type of Atrial Fibrillation [Count of Participants; unit: Participants]
  Paroxysmal | 66 | 65 | 131
  Persistent | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Time to First Event of Symptomatic Atrial Fibrillation/Atrial Flutter (AF/AFL) or All Cause Mortality (ACM) During the 24-week Follow-up Period After Establishment of Stable Sinus Rhythm (SR) on Study Drug [End of Treatment Week 24].
Description: Time-to-event is calculated as the date of the event minus the date of initiation of efficacy follow-up, with 1 added in order to include both the start date and end date of the interval. Cox's proportional hazards model will be used to calculate estimated hazard ratios and 95% confidence intervals. The calculations will be performed with the SAS PHREG procedure, with the stratification variables specified in the STRATA statement and the treatment group comparator and any covariates being examined specified in the MODEL statement. For the primary endpoint, the appropriateness of assuming proportional hazards will be explored by the graphing of log (-log(survival function)) over follow-up for each treatment group.
Time Frame: end of treatment week 24
Population: Time to first event of symptomatic atrial fibrillation/atrial flutter (AF/AFL) or all cause mortality (ACM) during the 24-week Follow-up Period after establishment of stable sinus rhythm (SR) on study drug [end of treatment week 24]. Results from participants were combined for analysis within each treatment arm. Mean time to event (days) is presented for the participants experiencing an event.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
Number analyzed (Participants) | 69 | 67
days | 35.9 [9 to 53] | 33.2 [6 to 47]
Statistical Analysis 1: Comparison: Bucindolol Hydrochloride vs Metoprolol Succinate; Test type: Superiority; p = 0.905, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [.72 to 1.45]

2. Secondary Outcome: Time to First Event of Symptomatic or Asymptomatic AF/AFL or ACM During the 24-week Follow-up Period After Establishment of Stable SR on Study Drug [End of Treatment Week 24]
Description: Number of days on study medication before participant experienced symptomatic or asymptomatic atrial fibrillation, atrial flutter, or all-cause mortality during the 24 week follow up period.
Time Frame: end of treatment week 24
Population: Time to first event of symptomatic or asymptomatic atrial fibrillation/atrial flutter (AF/AFL) or all cause mortality (ACM) during the 24-week Follow-up Period after establishment of stable sinus rhythm (SR) on study drug [end of treatment week 24]. Mean time to event (days) is presented for the participants experiencing an event.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
Number analyzed (Participants) | 73 | 70
days | 37.86 [9 to 53] | 31.06 [6 to 40.5]
Statistical Analysis 1: Comparison: Bucindolol Hydrochloride vs Metoprolol Succinate; Test type: Superiority; p = 0.961, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.71 to 1.42]

3. Secondary Outcome: Number of Patients With Adequate Ventricular Rate Control During the 24-week Follow-up Period
Description: Number of patients with adequate ventricular rate control following the start of medication during the 24-week Follow-up Period
Time Frame: end of treatment week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
Number analyzed (Participants) | 134 | 133
Participants | 84 | 116

4. Secondary Outcome: Total Number of Hospitalization Days Per Patient (All-cause) During the Total Study Period (24 Weeks)
Description: Total number of hospitalization days per patient (all-cause) following the start of study medication during the Total Study Period (24 weeks). Hospitalization was defined by a hospital admission (note that same day admit and discharge equates to 0 days duration), ER visits were not counted as events.
Time Frame: 24 weeks
Population: A summary of all-cause and HF hospitalizations by treatment group over the 24-week study period
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Unique Inpatient Hospitalizations
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
Number analyzed (Participants) | 60 | 51
Number analyzed (Unique Inpatient Hospitalizations) | 123 | 87
days | 2 [1 to 4] | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: Results were collected from first dose of study drug to the later of 30 days after last dose or last study evaluation (final visit) for each participant ("total study period"; e.g., up to day 1184). Adverse Events were not collected per specific doses, rather participants were combined for analysis within each treatment arm. All AEs reported during the course of the study were coded to a body system and preferred term using the Medical Dictionary for Regulatory Activities (medDRA) version 6.1.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Bucindolol Hydrochloride: bucindolol hydrochloride (bucindolol)
  Capsules were available in the following dosage strengths to be taken twice daily (with or without food): 6.25mg, 12.5mg, 25mg, 50mg, and 100mg.
  bucindolol hydrochloride
- Metoprolol Succinate: metoprolol succinate (Toprol-XL)
  Capsules were available in the following dosage strengths to be taken twice daily (with or without food): 25mg, 50mg, 100mg, 200mg and/or matching placebo oral capsule to maintain blinded dosing.
  metoprolol succinate
  Placebo oral capsule
Arm/Group | Bucindolol Hydrochloride | Metoprolol Succinate
All-Cause Mortality (participants affected / at risk) | 3/134 | 3/133
Serious Adverse Events (participants affected / at risk) | 33/134 | 26/133
Other Adverse Events (participants affected / at risk) | 100/134 | 95/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bucindolol Hydrochloride (N=134) | Metoprolol Succinate (N=133)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 7 (7)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylcoccal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic necrotic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1) | 1 (1)
Device lead damage (Product Issues) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vascular stent restenosis (General disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bucindolol Hydrochloride (N=134) | Metoprolol Succinate (N=133)
Cardiac failure congestive (Cardiac disorders) | 8 (8) | 10 (10)
Bradycardia (Cardiac disorders) | 5 (5) | 9 (9)
Cardiac failure (Cardiac disorders) | 7 (7) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 6 (6)
Constipation (Gastrointestinal disorders) | 8 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5) | 6 (6)
Hypotension (Vascular disorders) | 13 (13) | 10 (10)
Fatigue (General disorders) | 6 (6) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Metabolism and nutrition (Metabolism and nutrition disorders) | 19 (19) | 16 (16)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Investigations (Investigations) | 17 (17) | 10 (10)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 6 (6)
Psychiatric disorder (Psychiatric disorders) | 2 (2) | 12 (12)
Eye disorder (Eye disorders) | 8 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 13 (13) | 8 (8)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT01970501/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT01970501/SAP_001.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT01970501/ICF_002.pdf